CLINICAL TRIAL: NCT00645203
Title: An Open-Label, Safety and Efficacy Study of Cefdinir Oral Suspension, 25 mg/kg Once Daily, in Pediatric Subjects With Acute Otitis Media
Brief Title: Safety and Efficacy Study of Cefdinir Oral Suspension, in Pediatric Subjects to Treat Acute Otitis Media
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Angela M Nilius, Ph.D., Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M01-352
Record Dates: First submitted 2008-03-20; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Cefdinir

ARMS (1):
- 1 (Other)
  Interventions: Drug: cefdinir

INTERVENTIONS:
Drug: cefdinir — cefdinir oral suspension, 25 mg/kg once daily for 10 days
  Other Names: ABT-198, Omnicef, cefdinir

SUMMARY:
To evaluate the safety and efficacy of cefdinir oral suspension in children between 6 months and 4 years of age, with acute otitis media, who are at risk of persistent or recurrent otitis media.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children between 6 months and 4 years of age
* Weight does not exceed 40 kg
* Clinical diagnosis is acute otitis media
* Have evidence of middle ear fluid
* At risk for persistent or recurrent otitis media
* Generally in good health

Exclusion Criteria:

* Sensitivity or allergy to penicillins or cephalosporins or inability to take oral medications
* Presence of tympanostomy tubes, ventilation tube or perforated tympanic membrane, in either ear
* Treatment with any anti-infective agent within 3 days prior to the study or treatment with a long-acting injectable antimicrobial agent (e.g. , penicillin G benzathine) within 4 weeks prior to the study
* Concomitant infection, that requires additional antimicrobial therapy
* Presence of a disease, complicating factor (e.g., mastoiditis), or structural abnormality that would preclude evaluation of the patient's therapeutic response

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 447 (Actual)
Dates: Start 2002-07; Primary Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Bacteriological Response | 30 days
Clinical response | 30 days
Change in the otoscopic findings | 30 days

SECONDARY OUTCOMES:
Physical exam; Vital signs; Use of concomitant medications | 59 days
Adverse events assessment | 45 days with follow-up to a satisfactory conclusion
Laboratory evaluations | 30 days

CONTACTS AND LOCATIONS:
Locations (20):
- United States (12):
  - Scottsdale, Arizona
  - Clovis, California
  - Dinuba, California
  - Folsom, California
  - Denver, Colorado
  - Brooklyn, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Erie, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Salt Lake City, Utah
- Chile (2):
  - Providencia, Santiago Metropolitan
  - Puente Alto, Santiago
- Costa Rica (2):
  - Uruca, Provincia de San José
  - San José
- Santo Domingo, Dominican Republic
- Guatemala City, Guatemala
- Beersheba, Israel
- Panama City, Panama